CLINICAL TRIAL: NCT05884281
Title: Efficacy of Roflumilast in Prevention of Peripheral Neuropathy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Noha Mansour, Principal investigator-Lecturer of Clinical Pharmacy-Clinical Pharmacy and Pharmacy Practice Department, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 8/2023
Record Dates: First submitted 2023-05-22; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Peripheral Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator)
  Interventions: Drug: Roflumilast
- Control (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Roflumilast — 0.5 mg once daily for treatment period
  Arms: Intervention
Drug: Placebo — Placebo for treatment period
  Arms: Control

SUMMARY:
There are several mechanisms concerning pathophysiology of paclitaxel induced peripheral neuropathy. One of the main mechanisms is induction of Schwann cell dedifferentiation by paclitaxel. At the preclinical level, roflumilast potently inhibited paclitaxel-induced dedifferentiation of cultured Schwann cells, yet this positive effect have not been clinically investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Breast cancer patients who will receive paclitaxel post-anthracycline therapy.
2. Eastern Cooperative Oncology Group (ECOG) performance status from 0 to 2.
3. Adequate bone marrow function (white blood count ≥4,000/mm3, platelet count≥100,000/mm3), liver function (serum total bilirubin <1.5 mg/dl), renal function (creatinine < 1.5 mg/dl).

Exclusion Criteria:

1. Patients with signs and symptoms of clinical neuropathy at baseline.
2. Patients with diabetes mellitus or alcoholic disease.
3. Patients receiving vitamin/ supplementation drugs that interfere with the study intervention.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of chemotherapy induced-peripheral neuropathy using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) criteria | 8 weeks post intervention
  Number of patients reported neuropathy from paclitaxel

IPD SHARING:
Plan to Share IPD: Undecided